CLINICAL TRIAL: NCT04110392
Title: Effect of Consumption of a Beverage of Chaya (Cnidoscolus Chayamansa) on Lipid Concentration, Lipid Peroxidation and Antioxidant Status of Patients With Dyslipidemia
Brief Title: Effect of Consumption of Chaya on Lipid Concentration and Antioxidant Status of Patients With Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad de la Península de Yucatán (Other)
Responsible Party: Principal Investigator, Azalia Avila Nava, PhD, Researcher in medical sciences, Hospital Regional de Alta Especialidad de la Península de Yucatán
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-030
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: It is quasi-experimental and it was proposed before and after study, the study will be consisting of a pre-visit, 6 subsequent visits and a last visit to deliver results to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chaya (Cnidoscolus chayamansa) (Experimental): Chaya Water Beverage of Chaya will be prepared as follows: 40 g of Chaya leaves will be treated with a commercial brand disinfectant following the manufacturer's instructions for use, then added 1L of purified water and mixed in blender. Finally, 500 mL of it will be placed in bottles. Participants will be instructed to consume 1 bottle per day for 6 weeks. 7 bottles will be delivered at each visit, which will be consumed during the week; participants will be instructed to keep the water refrigerated until it is consumed.
  Interventions: Dietary Supplement: Chaya (Cnidoscolus chayamansa)

INTERVENTIONS:
Dietary Supplement: Chaya (Cnidoscolus chayamansa) — Chaya Water Beverage of Chaya will be prepared as follows: 40 g of Chaya leaves will be treated with a commercial brand disinfectant following the manufacturer's instructions for use, then added 1L of purified water and mixed in blender. Finally, 500 mL of it will be placed in bottles. Participants will be instructed to consume 1 bottle per day for 6 weeks. 7 bottles will be delivered at each visit, which will be consumed during the week; participants will be instructed to keep the water refrigerated until it is consumed.

SUMMARY:
Currently, the changes generated in lifestyle, such as excessive consumption of saturated fats and refined carbohydrates, as well as the decrease in the intake of fiber, fruits, vegetables and antioxidants, as well as physical inactivity, have generated an increase in the prevalence of dyslipidemias. Dyslipidemias are a disorder of blood lipid and lipoprotein concentration, which increases the risk of developing atherosclerosis and cardiovascular diseases. In Mexico, the dyslipidemias are present in one in four Mexicans over 20 years old. However, in Yucatan increases this frequency increases due to one in three people suffer from dyslipidemia. Its prevalence is even higher in overweight subjects, diabetes and high blood pressure. Thus, it is important to search for strategies to reduce dyslipidemias, as well as the complications associated with them. The treatment and prevention of dyslipidemia is through dietary treatment, which may be accompanied by the consumption of foods that generate beneficial health effects due to the presence of bioactive compounds. Chaya (Cnidoscolus chayamansa) is a plant use in popular medicine to treat medicine in the treatment of chronic degenerative diseases. It contained different bioactive compounds such as flavonoids, vitamin C and polyphenols such as quercetin and kaempferol. Compounds that have been assigned various beneficial effects such as decreased triglyceride concentrations, cholesterol, malondialdehyde, C-Reactive protein, oxidized LDL, which are alterations that are present in dyslipidemia. Therefore, the consumption of this food could be an adequate strategy for subjects with dyslipidemia in Yucatan and Mexico due to the anti-inflammatory and antioxidant effects, and could reduce the risk of developing atherosclerosis and cardiovascular diseases.

DETAILED DESCRIPTION:
The protocol will be carried out in the Hospital Regional de Alta Especialidad de la Península de Yucatán (HRAEPY). It is quasi-experimental and it was proposed before and after study, the study will be consisting in 6 subsequent visits and a last visit to deliver results to the participant.

In the pre-visit, the subjects will be evaluated to determine if they meet the inclusion criteria. They will be explained what the study consists of, the characteristics, the risks and the expected benefits after the intervention, they will be asked to read the consent letter, doubts will be clarified about it and if the participant agrees to be in the study the signature will be made of the consent letter.

At the beginning and end will be taken two blood samples of 5 mL to each participant. One will be to obtain the serum and measure cholesterol-HDL, cholesterol-LDL, triglycerides, total cholesterol, glucose, antioxidant activity, malondialdehyde (MDA) and C-reactive protein. The second sample will be to the extraction of peripheral leukocyte blood mononuclear cells and determine the gene expression of antioxidants enzymes superoxide dismutase (SOD) and catalase (CAT). Blood pressure will be measured with a digital baumanometer while the participant will remain seated with the right arm uncovered. The measurement will be carried out 6 times, in intervals of 3 minutes. The first measurement will be discarded and the average of the remaining measurements will be reported. In the visits will bring to each participant an attachment to reported intake of the beverage. During the following ones it will always be questioned if there is any problem with the drinking the beverage of Chaya.

At the end of the study, participants will be given the document with their results and will be given recommendations for weight control, dietary recommendations to improve lipid concentrations. They will refer to their doctor for follow-up with their laboratory results for their control.

Description of the intervention

Chaya Water Beverage of Chaya will be prepared as follows: 40 g of Chaya leaves will be treated with a commercial brand disinfectant following the manufacturer's instructions for use, then added 1L of purified water and mixed in blender. Finally, 500 mL of it will be placed in bottles. Participants will be instructed to consume 1 bottle per day for 6 weeks. 7 bottles will be delivered at each visit, which will be consumed during the week; participants will be instructed to keep the water refrigerated until it is consumed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female.
* Adults between 20 and 60 years.
* BMI ≥ 20 and ≤ 39.9 kg / m².
* Mestizo Mexicans: parents and grandparents born in Mexico.
* Patients diagnosed with dyslipidemia.
* Dyslipidemia will be defined by any? alteration in the concentrations of the following lipoproteins: LDL cholesterol> 130mg/dL or total cholesterol> 200 mg/dL or triglycerides> 150 mg/dL
* Patients should know how to read and write.
* Signature of informed consent.

Exclusion Criteria:

* Patients with any type of diabetes previously diagnosed
* Patients with acquired diseases that produce secondary obesity and diabetes.
* Patients who have suffered a cardiovascular event.
* Weight loss> 3 kg in the last 3 months.
* Catabolic diseases such as cancer and acquired immunodeficiency syndrome.
* Positive smoking.
* Drug treatment:

  * Antihypertensive drugs (thiacyclic, loop or potassium-sparing diuretics, angiotensin II receptor blockers, alpha blockers, calcium antagonists, beta blockers).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline triglycerides concentration at 6 weeks of intervention | At the beginning of the study and after 6 weeks of intervention
  Serum triglyceride measurement by the method of colorimetry enzymatic
Change from baseline Lipoproteins concentration at 6 weeks of intervention | At the beginning of the study and after 6 weeks of intervention
  Total cholesterol, LDL and HDL measurement by the method of colorimetry enzymatic

SECONDARY OUTCOMES:
Change from baseline blood gene expression of superoxide dismutase at 6 weeks of intervention | At the beginning of the study and after 6 weeks of intervention
  Gene expression of superoxide dismutase measurement by qPCR method
Change from baseline blood gene expression of catalase at 6 weeks of intervention | At the beginning of the study and after 6 weeks of intervention
  Blood gene expression of catalase measurement by quantitative polymerase chain reaction (qPCR) method
Change from baseline serum antioxidant activity at 6 weeks of intervention | At the beginning of the study and after 6 weeks of intervention
  Serum antioxidant activity measurement by spectrophotometric method
Change from baseline serum C-Reactive Protein at 6 weeks of intervention | At the beginning of the study and after 6 weeks of intervention
  Serum C-Reactive Protein measurement by the method of colorimetry enzymatic

CONTACTS AND LOCATIONS:
Overall Officials: Azalia Avila Nava, PhD, Principal Investigator — Hospital Regional de Alta Especialidad de la Península de Yucatán
Locations (1):
- Hospital Regional de Alta Especialidad de la Península de Yucatán, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Rodriguez RV, Gutierrez-Rebolledo GA, Mendez-Bolaina E, Sanchez-Medina A, Maldonado-Saavedra O, Dominguez-Ortiz MA, Vazquez-Hernandez M, Munoz-Muniz OD, Cruz-Sanchez JS. Cnidoscolus chayamansa Mc Vaugh, an important antioxidant, anti-inflammatory and cardioprotective plant used in Mexico. J Ethnopharmacol. 2014 Feb 3;151(2):937-43. doi: 10.1016/j.jep.2013.12.004. Epub 2013 Dec 11. PMID 24333962
- [Background] Loarca-Pina G, Mendoza S, Ramos-Gomez M, Reynoso R. Antioxidant, antimutagenic, and antidiabetic activities of edible leaves from Cnidoscolus chayamansa Mc. Vaugh. J Food Sci. 2010 Mar;75(2):H68-72. doi: 10.1111/j.1750-3841.2009.01505.x. PMID 20492237
- [Background] Kuti JO, Kuti HO. Proximate composition and mineral content of two edible species of Cnidoscolus (tree spinach). Plant Foods Hum Nutr. 1999;53(4):275-83. doi: 10.1023/a:1008081501857. PMID 10540979